CLINICAL TRIAL: NCT05124106
Title: In Vivo Proof-of-principle Study of Raman Spectroscopy in Trial Participants With Bladder Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Proff Dr Jürgen Popp, Leibniz Institute, IPHT, Jena, Germany (Unknown); Karin Mogensen urologist, Herlev hospital, Copenhagen, Denmark (Unknown); Proff Dr Iwan Schie, Leibniz Institute, IPHT, Jena, Germany (Unknown)
Responsible Party: Principal Investigator, Gregers Gautier Hermann, Consultant Urologist, University Hospital Bispebjerg and Frederiksberg
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Clinical Protocol (MIB)
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Endoscopic Bladder Cancer Diagnosis With Raman
Keywords: Bladder cancer; Raman spectrometry; In vivo diagnostics
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: Tumor identified during endoscopy of the bladder is examined with Raman spectrometry. Tumor is resected. Histopathological diagnosis is compared with results of Raman spectrometry.
Masking Description: Patient tumor stage is unknown for the examiner.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic ability of Raman spectrometry (Experimental): Endoscopic Raman spectrometry during endoscopic bladder cancer surgery
  Interventions: Diagnostic Test: Raman Spectrometry

INTERVENTIONS:
Diagnostic Test: Raman Spectrometry — Bladder tumor is examined with Raman spectrometry during endoscopy

SUMMARY:
The purpose with this clinical investigation is to perform Raman spectroscopy inside the vivid bladder and to acquire Raman spectra of normal and tumour bladder tissue, and in a post-processing step to determine the grade of the tumor.

DETAILED DESCRIPTION:
The purpose with this clinical investigation is to perform Raman spectroscopy inside the vivid bladder and to acquire Raman spectra of normal and tumour bladder tissue, and in a post-processing step to determine the grade of the bladder tumor.

The recordings and overall results will be compared to standard histo/cytopathological examination of urological tissue to achieve a clinical useful concordance between gold standard histo/cytopathological diagnosis and diagnostic information established by Raman.

The MIB RAMAN SYSTEM in combination with a Raman probe will be used in the operating theatre at Herlev/Copenhagen hospital urology department, where the rigid resectoscopes will be used while the trial participant is under general anesthesia. Each measurement takes about 1-5 seconds and the whole procedure with the fiber optic probes is expected to prolong the operation with 10-15 minutes.

ELIGIBILITY:
Inclusion Criteria:

After booking for surgery the trial participants will be informed orally about the study and written material will be given by a doctor or nurse form the study group. If the trial participant accept to enter the study, written informed consent will be obtained. The trial participant will be informed that they can withdraw the informed consent at any time and the treatment will be according to the guidelines of the department.

Exclusion Criteria:

* Macroscopic hematuria
* Pregnant or breast-feeding women
* Expected poor compliance
* Persons < 18 years
* Persons who do not read or understand Danish
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of tumor grade by Raman spectometry | 4 weeks
  To achieve a clinical useful concordance between gold standard histo/cytopathological diagnosis and the information provided through Raman spectroscopy.

SECONDARY OUTCOMES:
To evaluate feasibility of handling the diagnostic optic equipment (MIB RAMAN SYSTEM), the Raman probe and the software, when the urologist examines the bladder for lesions. | 4 weeks
  Examine results on the sensitivity and specificity for "diagnosis" (normal tissue/tumour) in 30 trial participants using the developed MIB RAMAN SYSTEM.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev hospital, Urology department, Herlev, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No